CLINICAL TRIAL: NCT01728571
Title: LungVITamin D and OmegA-3 Trial
Brief Title: LungVITamin D and OmegA-3 Trial (lungVITAL)
Acronym: lungVITAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard School of Public Health (HSPH) (Other)
Responsible Party: Principal Investigator, Diane Gold, Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: 2010-P-000622
Record Dates: First submitted 2012-10-25; First posted 2012-11-20 (Estimated); Last update posted 2025-02-06 (Actual); Status verified 2024-08

CONDITIONS: COPD; Asthma; Pulmonary Function; Pneumonia
Keywords: COPD; asthma; pulmonary function; pneumonia
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Asthma; Pneumonia | interventions — Cholecalciferol; Fish Oils; Omacor; Eicosapentaenoic Acid; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Vitamin D3 + fish oil (Active Comparator): Dietary Supplement: vitamin D3 Drug: omega-3 fatty acids (fish oil)
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: fish oil
- Vitamin D3 + fish oil placebo (Active Comparator): Dietary Supplement: vitamin D3 Dietary Supplement: fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3; Dietary Supplement: Fish oil placebo
- Vitamin D3 placebo + fish oil (Active Comparator): Drug: omega-3 fatty acids (fish oil) Dietary Supplement: vitamin D3 placebo
  Interventions: Dietary Supplement: fish oil; Dietary Supplement: Vitamin D3 placebo
- Vitamin D3 placebo + fish oil placebo (Placebo Comparator): Dietary Supplement: vitamin D3 placebo Dietary Supplement: fish oil placebo
  Interventions: Dietary Supplement: Vitamin D3 placebo; Dietary Supplement: Fish oil placebo

INTERVENTIONS:
Dietary Supplement: Vitamin D3
  Other Names: Vitamin D3 (cholecalciferol), 2000 IU per day. Other Name: cholecalciferol
  Arms: Vitamin D3 + fish oil; Vitamin D3 + fish oil placebo
Dietary Supplement: fish oil
  Other Names: Omacor; 1 g per day as a fish oil capsule, containing 840 milligrams of marine omega-3 fatty acids (460 mg of eicosapentaenoic acid [EPA] and 380 mg of docosahexaenoic acid [DHA]).
  Arms: Vitamin D3 + fish oil; Vitamin D3 placebo + fish oil
Dietary Supplement: Vitamin D3 placebo
  Arms: Vitamin D3 placebo + fish oil; Vitamin D3 placebo + fish oil placebo
Dietary Supplement: Fish oil placebo
  Arms: Vitamin D3 + fish oil placebo; Vitamin D3 placebo + fish oil placebo

SUMMARY:
The VITamin D and OmegA-3 TriaL (VITAL; NCT 01169259) is an ongoing randomized clinical trial in 25,871 U.S. men and women investigating whether taking daily dietary supplements of vitamin D3 (2000 IU) or omega-3 fatty acids (Omacor® fish oil, 1 gram) reduces the risk of developing cancer, heart disease, and stroke in people who do not have a prior history of these illnesses.

This ancillary study is being conducted among participants in VITAL and will examine whether vitamin D or fish oil reduces respiratory morbidity, including COPD and asthma exacerbations, the risk of pneumonia, and airflow obstruction/decline of pulmonary function; and whether either of these interventions improves asthma control.

DETAILED DESCRIPTION:
Chronic obstructive lung disease (COPD) and pneumonia are leading causes of death in United States and worldwide. COPD, which is also a significant source of disability, is increasing in prevalence. Approximately 14 million adults have asthma, which leads to approximately 12 million missed work days per year in the United States. In adults, COPD and asthma often coexist. Treatment options for COPD are limited, and prevalence of vitamin D deficiency is high. COPD lung disease (COPD, asthma, airflow obstruction), and most COPD additional co-morbidities responsible for COPD progression (e.g., respiratory infections/pneumonia, muscle weakness, cardiac failure) may benefit from vitamin D supplementation therapy, but this requires rigorous testing. Marine omega-3 fatty acids work through different pathways from vitamin D to affect inflammation. Observational studies and clinical trials suggest that consumption of fish and/or fish oil may protect against COPD, asthma or pneumonia, but the data are not consistent. Thus, there is a compelling need for a clinical trial to evaluate the potential benefits or risks of vitamin D and fish oil supplementation on COPD and asthma exacerbations, airflow obstruction and decline of lung function, and risk of pneumonia.

The primary outcomes of interest in Lung VITAL are COPD exacerbations; airflow obstruction and decline of pulmonary function; and pneumonia. Asthma exacerbations and asthma control are secondary outcomes. A tertiary goal is to assess whether the effects of the interventions differ by baseline dietary intake or baseline blood levels of the nutrients.

Depending on the primary outcome, Lung VITAL will be conducted among all participants in VITAL (NCT 01169259), or in subsets of the VITAL population who were followed by detailed respiratory questionnaire and/or lung function testing.

ELIGIBILITY:
* This study is open to all VITAL participants (NCT 01169259). Population includes men 50 years of age or older and women 55 years of age or older in the United States
* Participants who live in selected metropolitan areas of the U.S. (where we set up the infrastructure for clinic or home visits), are eligible for pulmonary function measurements.

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25871 (Actual)
Dates: Start 2010-07; Primary Completion 2018-11-10 (Actual); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
COPD exacerbations in the past year over the course of the study | at baseline (before randomization), 1-year, 2-year, 3-year,4-year, 5-year
  Baseline respiratory symptom status, respiratory disease diagnoses, and COPD (chronic obstructive pulmonary disease) exacerbations in the past year are measured pre-randomization and annually during follow-up.
Airflow obstruction/change in pulmonary function | pre-randomization and after 2 years follow-up
  In a sub-group of study participants pulmonary function will be measured pre-randomization and after 2 years of follow-up
Pneumonia in the past year over the course of the study | at baseline (before randomization), 1-year, 2-year, 3-year,4-year, 5-year
  Pneumonia in the past year (overall and in those with COPD and asthma) is measured pre-randomization and annually during follow-up.

SECONDARY OUTCOMES:
Asthma exacerbations and asthma control in the past year over the course of the study | at baseline (before randomization), 1-year, 2-year, 3-year,4-year, 5-year
  Participants who report an asthma diagnosis are asked questions related to respiratory illness exacerbations and asthma control annually during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Diane R Gold, MD, MPH, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Gold DR, Carey VJ, Hersh CP, Wan E, Camargo CA Jr, Lee IM, Cook NR, Nassikas N, Buring JE, Manson JE, Luttmann-Gibson H. Vitamin D Supplementation, Chronic Obstructive Lung Disease and Asthma Exacerbations, and Lung Function Decline. J Nutr. 2025 May;155(5):1417-1428. doi: 10.1016/j.tjnut.2025.02.003. Epub 2025 Feb 6. PMID 39922497
- [Derived] Gold DR, Litonjua AA, Carey VJ, Manson JE, Buring JE, Lee IM, Gordon D, Walter J, Friedenberg G, Hankinson JL, Copeland T, Luttmann-Gibson H. Lung VITAL: Rationale, design, and baseline characteristics of an ancillary study evaluating the effects of vitamin D and/or marine omega-3 fatty acid supplements on acute exacerbations of chronic respiratory disease, asthma control, pneumonia and lung function in adults. Contemp Clin Trials. 2016 Mar;47:185-95. doi: 10.1016/j.cct.2016.01.003. Epub 2016 Jan 16. PMID 26784651